CLINICAL TRIAL: NCT03240718
Title: Randomized, Controlled, Within-patient, Single-blinded Pilot Study to Evaluate the Efficacy of the Ablative Fractional CO2 Laser in the Treatment of Hypertrophic Scars in Adult Burn Patients
Brief Title: Pilot Study of the Ablative Fractional CO2 Laser in Hypertrophic Scars in Adult Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE14-122
Record Dates: First submitted 2017-02-03; First posted 2017-08-07 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2015-12

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser treated HSc scar (Experimental): Co2 laser treatment
  Interventions: Procedure: Laser treatment
- Control scar (No Intervention): Standard care

INTERVENTIONS:
Procedure: Laser treatment — CORE fractional CO2 laser treatment
  Arms: Laser treated HSc scar

SUMMARY:
This is a randomized, controlled, within-patient, single-blinded, pilot study that will evaluate the impact of laser treatment on burn HSc relative to self-matched control scars. The studied primary outcomes of treatment are scar pliability, thickness, vascularity, pain, itch and patient satisfaction.

DETAILED DESCRIPTION:
Prior to treatment initiation, two independent scars sites will be selected and an anatomically- on each individual. At the selected treatment site the scar will be treated with the CORE fractional CO2 laser Participants will receive 3 treatment sessions scheduled 4 weeks apart. The scar sites will be evaluated at baseline, immediately before the 3rd treatment and 12 weeks after their final treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type <IV (37),
* Have sustained a thermal burn injury,
* Have at least 2 independent sites that show clinical evidence of HSc,
* Are 2 months or more post-injury.

Exclusion Criteria:

* Subjects with skin phototypes IV or higher,
* With history of keloidal scarring,
* Who have coagulation disorder,
* Are taking immunosuppressive medications,
* If the mechanism of injury is an electrical, chemical, or cold injury,
* Any underlying active skin disease,
* Have taken oral Isotreinoin within the last 6 months,
* Photosensitivity or have taken photosensitizing medications,
* Pregnancy,
* Previous treatment with dermabrasion, chemical peel, laser or intense pulsed light treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Skin Characteristics changes | baseline, 12 weeks and 24 weeks
  Erythema, elasticity and thickness measures

SECONDARY OUTCOMES:
Satisfaction Questionnaire | baseline, 24 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Nedelec, PhD, Principal Investigator — CRCHUM

IPD SHARING:
Plan to Share IPD: Yes